CLINICAL TRIAL: NCT02841215
Title: A Randomized Controlled Double-blind Trial Assessing the Efficacy of a 400µg/kg Ivermectin /5% Permethrin / Emollient Cream Regimen in Patients With Crusted Scabies as Compared to a 200µg/kg Ivermectin /5% Permethrin /Emollient Cream Regimen
Brief Title: Efficacy Study Between Two Different Dosages of an Antiparasitic in Patients With Crusted Scabies
Acronym: GALECRUSTED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P140939
Record Dates: First submitted 2016-06-30; First posted 2016-07-22 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Gale; Severe Forms of Scabies; Oral Parasitic Drug; Ivermectin
Keywords: Gale; Severe forms of scabies; Oral parasitic drug; Ivermectin
MeSH Terms: conditions — Galactosemias | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral ivermectin 400 µg/kg (Experimental): Oral ivermectin 400 µg/kg + topical treatment (permethrin 5% cream) + emollient cream (Dexeryl® or other)
  Interventions: Drug: Ivermectin 400 µg/kg
- Oral ivermectin 200 µg/kg (Active Comparator): Oral ivermectin 200 µg/kg + topical treatment (permethrin 5% cream) + emollient cream (Dexeryl® or other)
  Interventions: Drug: Ivermectin 200 µg/kg

INTERVENTIONS:
Drug: Ivermectin 200 µg/kg — Oral ivermectin 200 µg/kg three times (D0, D7 and D14) + topical treatment (permethrin 5% cream) on skin, hair and genital organs (D0 and D7) + emollient cream (Dexeryl® or other) daily on skin (D0 to D28)
  Arms: Oral ivermectin 200 µg/kg
Drug: Ivermectin 400 µg/kg — Oral ivermectin 400 µg/kg three times (D0, D7 and D14) + topical treatment (permethrin 5% cream) on skin, hair and genital organs (D0 and D7) + emollient cream (Dexeryl® or other)daily on skin (D0 to D28)
  Arms: Oral ivermectin 400 µg/kg

SUMMARY:
Severe forms of scabies (crusted scabies and profuse scabies) require a specific treatment. Ivermectin is a recommended treatment in common forms of scabies and represents a promising treatment in crusted scabies in case reports. However, response to ivermectin remains variable among studies, and there is no consensus on the schemes to adopt (dosages and administrations). Ivermectin at 400 µg/kg has already been used, without showing toxicity (in head lice treatment in particular). Investigators propose to demonstrate that 400µg/kg ivermectin dosage will show better efficacy than a 200µg/kg in patients with severe forms of scabies (crusted and profuse).

ELIGIBILITY:
Inclusion Criteria:

Patients ≥ 18 years old, diagnosed with severe forms of scabies

1. clinical criteria : cutaneous lesions of scabies

   * crusted scabies: at least two sites of hyperkeratosis will define crusted scabies and/or
   * profuse scabies : spreading lesions with erythematous scaly eruption of the neck, face or trunk without hyperkeratosis
2. paraclinical criteria:

   * Positive parasitological test
   * and/or dermoscopic exam with signs of scabies

Effective contraception for women in age of pregnancy Written consent from patient or his/her legal representant, trustworthy person or family member Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant and/or breastfeeding women
* Intolerance to ivermectin or topical treatment (permethrin 5% cream) or emollient cream
* Use of anti parasitic drug (ivermectin or albendazole) within the past 7 days
* Abnormal liver test results: ALT and/or AST >3N within the past 7 days (within 6 months if no hepatic history)
* Participation in other biomedical drug research
* Patient deprived of freedom
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Rate of a successful treatment defined by : -Two negative parasitologic and/or two dermoscopic exams | Days 21+/-2 days
  Parasitologic and/or dermoscopic exams will be perform at days 18 +/-2days and at days 21+/-2 days
Rate of a successful treatment defined by : - A clinical response : disappearance of clinical active lesions | Days 28+/- 2 days

SECONDARY OUTCOMES:
Rate of adverse effects | Days 18 +/-2 days, Days 21+/-2 days and Days 28+/-2 days

CONTACTS AND LOCATIONS:
Overall Officials: Giao DO-PHAM, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/24069468